CLINICAL TRIAL: NCT05789290
Title: Use of a Hilotherm Cryocompression Device to Reduce the Skin Temperature of the Knee to the Therapeutic Range of 10-15℃: a Prospective Cohort Study
Brief Title: Skin Temperature Reduction With Hilotherm Device
Status: Withdrawn | Type: Observational
Why Stopped: Unable to procure device under investigation following change in circumstances
Sponsor: University of Winchester (Other)
Collaborators: Physiolab Technologies Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: HWB_REC_230131_Faulkner
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group: This group will receive a 30-minute cryocompression treatment to one knee using a Hilotherm device, which is set to circulate water through the cuff at a maintained temperature of 10℃. The Hilotherm device will be administered according to the manufacturer's guidelines and each participant will undergo this treatment once.
  Interventions: Device: Hilotherm cryocompression device

INTERVENTIONS:
Device: Hilotherm cryocompression device — An electronic device that is capable of circulating warm or cooled water at a user-selected temperature between 10-30℃. Water is circulated from a central unit, through a tube, to a cuff wrapped around the intended therapy area (the knee). A treatment lasts for 30-minutes, at which point the device is turned off and the cuff is removed from the limb of the user.

SUMMARY:
Cryotherapy after surgery is widely utilised and has numerous practical applications for post-operative rehabilitation. Previous research has suggested that during cold therapy, the skin temperature of the knee should be reduced to 10-15°C to maximise the therapeutic benefits of cooling while avoiding the risk of cold injuries such as nerve damage and frostbite. The temperature to which a cryocompression device should be set in order to achieve a skin temperature within the therapeutic range of 10-15°C is unknown. Furthermore, there is evidence to suggest that the temperature setting of the device does not equal that to which the skin is reduced. Therefore, it is not sufficient to assume that the temperature setting of a cryocompression device accurately reflects the achieved skin temperature. Modern cryotherapy devices mostly consist of some sort of cuff that can be wrapped around the knee, with a connecting tube to a central unit that supplies and circulates cold water to and from the cuff in order to cool the intended body part. The Hilotherm is one such device for use in this way, but its ability to reduce skin temperature to within the target therapeutic range is unknown. The aim of this study is to determine whether the Hilotherm device is capable of reducing skin temperature of the knee to within the 10-15℃ therapeutic range during a standard 30-minute treatment.

DETAILED DESCRIPTION:
This prospective randomised controlled trial will recruit healthy adult volunteers from a university population to participate. A power analysis demonstrated that a total of 30 participants would be required to achieve a power of 0.8 and alpha error probability of 0.05 for a small-medium effect size of f=0.2. All eligible participants will first be required to provide informed consent prior to their participation in the study. Once this has been obtained, participants will each attend a single testing session lasting no longer than 60 minutes. The height and mass of the participants will be measured during the testing session in order to calculate BMI, and participants' age and sex will be recorded for inclusion inclusion in the later data analysis.

Participants will be required to remain in a seated position with their leg in full extension and elevated, parallel to the floor, for the duration of the test. The leg that will be used for the study will be randomly selected for each participant. Skin temperature will be measured using a thermocouple, which will be attached with tape 20 mm distal to the patella. The Hilotherm device will then be attached to the leg of the participant and the test will begin. The device will be set to apply the lowest possible temperature (10℃ ) to the knee to allow for an assessment of the maximal capability of the device to be conducted.

The temperature of the skin will be measured using a k-type thermocouple attached to an infrared thermometer immediately prior to the application of a device, and then every 5 minutes for the duration of the test. The length of a test will be 30 minutes, in accordance with the manufacturers' instructions/recommendations for each device.

Upon completion of a test, the cuff will be removed. If the temperature of the skin has been reduced to within 10-15℃, skin temperature will continue to be monitored every 5 minutes after the cuff has been removed until it rises above 15℃, at which point the test will end. This will allow for the total time to be measured that skin temperature remains within the target therapeutic range as a result of a single application of the cryocompression device. If the skin temperature is not reduced to within 10-15℃ while the cuff is worn, then the test will end after the cuff is initially removed. Upon completion of the test, the temperature sensor will be removed from the leg of the participant; thus completing their participation in the test and the study.

The following measures will be recorded: skin temperature at each time point, minimum skin temperature achieved, time to achieve minimum skin temperature, length of time with skin temperature within therapeutic range of 10-15℃. After each test, participants will also be asked to respond to the following question using a 5-point Likert scale: "How comfortable did you find the treatment you just experienced?" The possible answers to this question will be: "Very comfortable, Comfortable, Neutral, Uncomfortable, Very uncomfortable". This will provide insight into differences in perception of the treatment, which could be relevant for the likelihood of protocol adherence by patients in clinical settings.

The data will be analysed to detect any differences during testing compared to baseline measures. All data will be first subjected to a Kolmogorov-Smirnov test to assess whether they are normally distributed. A repeated measures analysis of variance will be performed on all normally distributed data. A Friedman test will be performed on any data that are not normally distributed.

Risk to participants is deemed to be very low for this study as the device temperature setting that will be used is within the target therapeutic zone, which is known to be safe for use with individuals who are not ordinarily contraindicated for cold therapy application.

Participants have the right to withdraw themselves and any collected data from the study at any time during, and for the first 7 days after, their participation without having to give a reason. They also have the right to terminate a test session at any time. Testing shall also be terminated as a result of any adverse reactions that emerge. Adverse reactions (e.g. pain) to the testing protocol are not expected due to the low-risk nature of the study, however any that occur shall be recorded and monitored until things return to baseline/normal. In order to monitor any pain/discomfort that might occur, a Numerical Pain Rating Scale (0-10 scale) will be within sight of the participant at all times during testing: a test will be terminated if reported pain/discomfort exceeds 5/10, though none is expected. Any reported pain (or other adverse reactions) shall be stored along with the data collected for that participant. If a test is terminated for a reason that could be mitigated in future, participants will be offered the opportunity to repeat the test another day, should they wish to continue taking part in the study. If a test is terminated due to an adverse reaction that can not be mitigated in future, the participant (and any collect-ed data) will be thanked for their time and withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age

Exclusion Criteria:

* BMI >40 kg/m2
* History of nerve damage or sensory deficit in the lower limbs (including frostbite)
* Hypersensitivity to cold, including hives
* Active inflammation or pain of the knee
* History of thrombosis, embolism, or other conditions related to impaired peripheral circulation
* Suffering from diagnosed diabetes, multiple sclerosis, rheumatoid arthritis, spinal cord injury, cardio-vascular disease, hypertension, Raynaud disease, cryoglobulinemia, or haemoglobinuria
* Confirmed or suspected tissue infection, an unstable fracture, a skin condition, or a tumour in the treatment area
* Cognitive impairment or communication barriers where adjustments can not be reasonably made

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers recruited primarily from a university population. All individuals willing to participate will be screened according to the abovementioned inclusion/exclusion criteria, and will be recruited until 30 people have completed their participation in the study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Skin temperature | 60 minutes
  Skin temperature will be measured using a thermocouple positioned 20 mm distal to the patella. This sensor will be attached prior to the cryocompression device being applied, and will remain in place until the testing session is complete and skin temperature is >15℃. (The therapeutic skin temperature range for cryotherapy is thought to be 10-15℃). Temperature will be measured prior to the cryocompression device being applied; every 5 minutes during the test; and every 5 minutes after a test until the skin temperature reaches >15℃.

SECONDARY OUTCOMES:
Subjective comfort | 60 minutes
  After each test, participants will also be asked to respond to the following question using a 5-point Likert scale: "How comfortable did you find the treatment you just experienced?" The possible answers to this ques-tion will be: "Very comfortable, Comfortable, Neutral, Uncomfortable, Very uncomfortable". This will provide insight into differences in perception of the treatment, which could be relevant for the likelihood of protocol adherence by patients in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: James Faulkner, PhD, Principal Investigator — University of Winchester
Locations (1):
- University of Winchester, Physiology Laboratory, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only researchers directly involved with the data collection of the study will have access to individual participant data. Data will be anonymised prior to analysis and only group data will be presented within resultant manuscripts.

REFERENCES:
- [Background] Wilke B, Weiner RD. Postoperative cryotherapy: risks versus benefits of continuous-flow cryotherapy units. Clin Podiatr Med Surg. 2003 Apr;20(2):307-22. doi: 10.1016/S0891-8422(03)00009-0. PMID 12776983
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Fang L, Hung CH, Wu SL, Fang SH, Stocker J. The effects of cryotherapy in relieving postarthroscopy pain. J Clin Nurs. 2012 Mar;21(5-6):636-43. doi: 10.1111/j.1365-2702.2010.03531.x. Epub 2011 Feb 20. PMID 21332855
- [Background] Waterman B, Walker JJ, Swaims C, Shortt M, Todd MS, Machen SM, Owens BD. The efficacy of combined cryotherapy and compression compared with cryotherapy alone following anterior cruciate ligament reconstruction. J Knee Surg. 2012 May;25(2):155-60. doi: 10.1055/s-0031-1299650. PMID 22928433
- [Background] Bellon M, Michelet D, Carrara N, Vacher T, Gafsou B, Ilhareborde B, Mazda K, Ferrero E, Simon AL, Julien-Marsollier F, Dahmani S. Efficacy of the Game Ready(R) cooling device on postoperative analgesia after scoliosis surgery in children. Eur Spine J. 2019 Jun;28(6):1257-1264. doi: 10.1007/s00586-019-05886-6. Epub 2019 Jan 31. PMID 30847706
- [Background] Selfe J, Hardaker N, Whittaker J and Hayes C. An investigation into the effect on skin surface temperature of three cryotherapy modalities. Thermology International. 2009; 19(4): 121-126.